CLINICAL TRIAL: NCT00544362
Title: Neoadjuvant Treatment for Operable Esophageal Cancer With 5-fluorouracil, Cisplatin, and Cetuximab and Concurrent Radiotherapy: Phase I/II Study
Brief Title: Fluorouracil, Cisplatin, Cetuximab, and Radiation Therapy in Treating Patients With Esophageal Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564075; FFCD-0505; EU-20756; EUDRACT-2006-004770-27; MERCK-FFCD-0505
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant chemoradiotherapy (Experimental): Weekly cetuximab (400 mg/m2 one week before start of radiotherapy RT and 250 mg/m2 during radiotherapyRT), and 5 FU (500 mg/m2 per day D1-D4) combined with cisplatin CDDP (40 mg/m2 D1) on week 1 and 5
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: fluorouracil; Procedure: conventional surgery

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving fluorouracil and cisplatin together with cetuximab and radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of fluorouracil and cisplatin when given together with cetuximab and radiation therapy in treating patients with esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of fluorouracil and cisplatin when administered with cetuximab concurrently with esophageal radiotherapy. (Phase I)
* To determine the complete histological response rate (after surgical resection). (Phase II)

Secondary

* To determine progression-free survival and overall survival. (Phase II)
* To determine the rate of resection with negative margins (R0). (Phase II)
* To determine the overall tolerance to neoadjuvant therapy. (Phase II)
* To determine the postoperative morbidity and mortality. (Phase II)

OUTLINE: This is a multicenter study. This is a dose-escalation study of cisplatin and fluorouracil.

Patients receive cetuximab IV over 2 hours on day -7, then IV over 1 hour on days 1, 8, 15, 22, and 29. Patients also receive cisplatin IV over 1 hour on day 1 or 2 and fluorouracil IV continuously on days 1-4, 8-11, 15-18, 22-25, and 29-32. Patients undergo radiotherapy 5 days a week for 5 weeks, beginning on day 1 of chemotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery within 6-8 weeks after completion of chemoradiotherapy.

After completion of study therapy, patients are followed at 1 month, every 4 months for 2 years, and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed epidermoid or glandular carcinoma of the thoracic esophagus

  * Invasive disease
  * Only Siewert type I gastroesophageal carcinoma allowed
* Resectable disease

  * T1N+, T2N0, T2N+, T3N0, or T3N+ (stage II or III)
  * No visceral metastases or mediastinal extensions compromising resectability

Exclusion criteria:

* Inoperable disease
* Invasion of the tracheo-bronchial tree
* Recurring esophageal paralysis
* Esopho-tracheal fistula
* Cervical esophageal carcinoma (< 19 cm above the dental arches)
* Multifocal esophageal carcinoma
* Superficial esophageal carcinoma (T1N0)
* Esophageal carcinoma in the lymph nodes that cannot be included in the radiotherapy field or cannot be completely surgically resected
* Proven metastatic disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-1
* Weight loss < 15%
* Absolute neutrophil count ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Creatinine ≤ 1.25 times upper limit of normal
* PTT ≥ 80%
* Albumin ≥ 35 g/L
* FEV1 > 1 L
* Not pregnant or nursing
* Fertile patients of must use effective contraception

Exclusion criteria:

* Known liver cirrhosis
* Renal insufficiency
* Respiratory insufficiency (i.e., severe dyspnea at rest or oxygen dependence)
* Progressive coronary insufficiency
* Myocardial infarction in the past 6 months
* Legally incapacitated
* Impossible to receive study therapy due to geographical, social, or psychological reasons
* Noncompliant within constraints of the study
* Hematologic malignancy or other cancer except carcinoma in situ of the uterine cervix, treated nonmelanoma skin cancer, or intramucous disease treated within the past 3 years

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior anticancer chemotherapy or radiotherapy
* Treatment with endoprosthesis
* Surgery (esophagectomy) planned without thoracotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Complete histologic response | After Surgery
Tolerance to neoadjuvant therapy | From Inclusion

SECONDARY OUTCOMES:
Progression-free and overall survival | From inclusion
Mortality | From Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Martina Schneider, Study Chair — Federation Francophone de Cancerologie Digestive
Locations (13):
- France (13):
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - C.H.U. de Brest, Brest
  - CHR Clermont Ferrand, Hotel Dieu, Clermont-Ferrand
  - Hopital Du Bocage, Dijon
  - Federation Francophone de Cancerologie Digestive, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospital Universitaire Hop Huriez, Lille
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Regional de Purpan, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy